CLINICAL TRIAL: NCT03741504
Title: Biological Anchorage With Selective Micro-osteroperforations (MOPs) in Canine Distalization
Brief Title: Biological Anchorage With Selective Micro-osteoperforations (MOPs) in Canine Distalization
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The requiered sample were not recruited due to COVID-19 pandemic
Sponsor: Fundación Universitaria CIEO (Other)
Collaborators: Universidad de Antioquia (Other)
Responsible Party: Principal Investigator, Sonia Patricia Plaza, Research coordinator Orthodontic Department, Fundación Universitaria CIEO
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 042
Record Dates: First submitted 2018-11-06; First posted 2018-11-15 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Teeth Mesial Drift; Bone Injury; Orthodontic Pathological Resorption of External Root
MeSH Terms: conditions — Mesial Movement of Teeth

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No micro-osteoperforations (No MOPs) (No Intervention): Canine Distalization without micro-osteoperforations Distalization of the upper canine in working phase with coil spring of 100 gr of force
- Micro-osteoperforations (MOPs) (Experimental): Canine Distalization with micro-osteoperforations at the start of the distalization Distalization of the upper canine in working phase with coil spring of 100 gr of force
  Interventions: Procedure: micro-osteoperforations (MOPs)

INTERVENTIONS:
Procedure: micro-osteoperforations (MOPs) — three (3) micro-osteoperforations (MOPs) in the cortical and medullar bone, distal to the upper canine. These MOPs will be at the apical, medial and gingival zone of the bone located at the distal surface of the canine in the buccal and in the palatal side. The deep of the MOPs will be at 6 mm. It is going to be done with a PROPEL
  Arms: Micro-osteoperforations (MOPs)

SUMMARY:
To evaluate the effect of selective micro-osteoperforations (MOPs) on the amount of distal movement of the upper canine, the mesio-distal inclination of the canine and the messiah movement of the upper first molar.

Methods: Clinical trial with Split mouth design in 35 orthodontic patients with bilateral extraction of the upper first premolar, each upper canine will be randomly assigned to the intervention (MOP) or to the control side. Participants will be followed for 3 months and the investigators will take periapical radiographs, cast models and clinical measurements before and after canine retraction. The measurements will be taken by previously calibrated operators. The results are going to be determined and compared between sides, with the corresponding statistical tests and the results are going to be analyzed.

DETAILED DESCRIPTION:
PICO QUESTION: ¿Does the amount of distal orthodontic movement of the upper canine increase in the side with MOPs compared with the side without MOPs? Population: Orthodontic patients with bilateral extraction of the upper first premolar (Split mouth design trial) Intervention: Distal movement of the upper canine with Selective MOPs (distal to canine) in one hemi-arch Comparison: Distal movement of the upper canine without MOPs in the other hemi-arch Outcome: Canine and first molar movements

GENERAL AIM:

- To evaluate the effect of selective micro-osteoperforations (MOPs) on the amount of distal movement of the upper canine, the M-D inclination of the canine and the mesial movement of the upper first molar.

METHODS

OVERVIEW OF DESIGN Study Design: Randomized controlled clinical trial in split mouth design.

* Randomly assign upper canines in to 2 sides in a split mouth design study: one side to receive intervention (MOPs) and the other side as a control (without MOPs).
* Then follow both sides for three months
* Split mouth design method: The investigators are going to randomly assign to the patients' left or right sides, one side for the intervention and the other side for the control (to eliminate the possibility of selection bias).
* Blinding: It is not possible to blind participants and clinical staff, but the investigators are going to blind the operators who will perform the measurements and the data analysis (single-blinded).

The participants will be with orthodontic fixed appliances (MBT prescription slot 0.022 "x0.028", canine torque 0 °), with working arches 0.019 "x0.025" stainless steel and with bilateral extractions of the first upper premolars for 6 months or more. For this moment the crowding must be resolved and there must be a space of 3 or more millimeters between the canines and second premolars.

The 4 upper incisors will be consolidated with a 0.010 "stainless steel ligature below the arch to prevent opening of anterior spaces.

Observation:

* No transpalatal arch (TPA) will be used in any of the participants
* It is going to place a mini-implant in the palate for reference point before the start of the experiment PLANS FOR RECRUITMENT Patients of the Clinic University (UniCIEO) and Antioquia University POTENCIAL CONFOUNDING VARIABLES
* Age
* Sex
* Systemic diseases not reported by the participant

ELIGIBILITY:
Inclusion Criteria:

* Class I or Class II malocclusion, division 1 (ANB: 0º-5º) with maxillary canines completely erupted with the need for canine retraction.
* Patients in the working phase with MBT prescription, slot 0.022" who have undergone extractions of bilateral upper premolar with more than three months before the time of upper canine distalization and with open space between the canine and the second premolar greater or equal to 3 mm.
* Age range between 14-40 years.
* Probing depth less than 4 mm in the upper canine

Exclusion Criteria:

* Patients with systemic disease.
* Medicated patients (prolonged use of antibiotics, phenytoin, cyclosporine, anti-inflammatory drugs, corticosteroids, systemic steroids, and calcium channel blockers).
* Pregnancy.
* Poor oral hygiene evident in more than two visits.
* Overjet ≥ 6 mm
* SN-GoGn ≥ 38 °
* Radiographic evidence of moderate to severe bone loss.
* Subjects with active periodontal disease
* Patients who smoke.
* Individuals with inadequately treated endodontic problems in the study area.

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2021-03-09 (Actual); Study Completion 2021-03-09 (Actual)

PRIMARY OUTCOMES:
Amount of distal movement of the upper canine | Change from baseline at three months
  Distance from a tangent to a reference point in the palate (third palatal ruga) to the distal side of the upper canine (measured in digital models)
Inclination of the upper canine, second premolar and first molar | Change from baseline at three months
  The angle between the long axis of the clinical crown and the reference plane the occlusal plane.(measured in digital models)
Angulation of the upper canine, second premolar and first molar | Change from baseline at three months
  The long axis of the posterior buccal surface is going to be measured relative to the occlusal plane (measured in digital models)
Amount of mesial movement of upper first molar | Change from baseline at three months
  Distance from a tangent to a reference point in the palate (third palatal ruga) to the mesial side of the upper first molar (measured in digital models)

SECONDARY OUTCOMES:
Periodontal status | Change from baseline at three months
  It's going to be measured by clinical exam
Evaluation of the perception of pain by the patient: VAS | Change from baseline at three months
  Pain visual analogue scale (AVS) - from 0 to 10 points, Higher values represent more pain perception by the participant
Number of participants with postoperative inflammation and/or infection | Change from baseline at three months
  Inflammation, infection by clinical exam
Number of upper canines with external root resorption | Change from baseline at three months
  Periapical radiograph

CONTACTS AND LOCATIONS:
Locations (2):
- Colombia (2):
  - UniCIEO, Bogotá, DC
  - Universidad de Antioquia, Bogotá, DC

IPD SHARING:
Plan to Share IPD: No
Individual participant data is going to be share only for statistical analysis